CLINICAL TRIAL: NCT02533908
Title: Combination of Nitrous Oxide 70% With Fentanyl Intranasal for Procedural Analgosedation in Children: A Prospective, Randomized, Double-blind, Placebo-controlled, Monocentric Study
Brief Title: Combination of Nitrous Oxide 70% With Fentanyl Intranasal for Procedural Analgosedation in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fentanyl-2015
Record Dates: First submitted 2015-07-20; First posted 2015-08-27 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-10

CONDITIONS: Inhalation of Nitrous Oxide; Opioid Analgesic Adverse Reaction; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl intranasal (Active Comparator): Fentanyl Sintetica 0.1mg/2ml: 1.5ug/kilogram intranasal= 0.03ml/kg once
  Interventions: Drug: Fentanyl intranasal
- NaCl 0.9% intranasal (Placebo Comparator): NaCl 0.9% Sintetica 18mg/2ml: same dosage as fentanyl= 0.03ml/kg
  Interventions: Drug: NaCl 0.9% intranasal

INTERVENTIONS:
Drug: Fentanyl intranasal — fentanyl is applied intranasally with a MAD (mucosal atomization device) prior to the application of nitrous oxide 70% analgosedation
  Other Names: Fentanyl Sintetica
  Arms: Fentanyl intranasal
Drug: NaCl 0.9% intranasal — Placebo is applied intranasally with a MAD (mucosal atomization device) Prior to the application of nitrous oxide 70% analgosedation
  Other Names: NaCl 0.9% Sintetica
  Arms: NaCl 0.9% intranasal

SUMMARY:
This study analyzes the analgesic efficacy and adverse events of nitrous oxide 70% combined with basic analgetics compared to nitrous oxide 70% with fentanyl intranasal for analgosedation for short and painful procedures in children.

DETAILED DESCRIPTION:
Nitrous oxide 70% (N20 70%) combined with 30% oxygen meets many criteria of an ideal pain medication for procedural analgosedation in children. At the emergency department of the Children's Hospital of Zurich, Switzerland, N20 70% is regularly used for short and painful orthopaedic procedures, mostly for reduction of dislocated forearm or finger fractures. The analgesic efficacy of N20 70% still remains controversial. Therefore, all children who are eligible for N20 70% receive additionally either fentanyl or placebo intranasal and then their behavior, level of sedation and adverse events are measured during the painful procedure. The hypothesis is that a combination of N20 70% and fentanyl intranasal is not significant better than N20 70% combined with basic analgetics.

ELIGIBILITY:
Inclusion Criteria:

* indication for nitrous oxide 70% application
* boys/girls aged 2-16 years
* informed consent

Exclusion Criteria:

* due to language barrier no sufficient communication possible to explain the study
* incompatibility to Fentanyl Sintetica
* incompatibility to morphinomimetics

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 402 (Actual)
Dates: Start 2015-09-21; Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Analgesic efficacy of nitrous oxide 70% versus nitrous oxide 70% combined with fentanyl intranasal using the FLACC score | up to 18 months
  the Patient is videotaped during the painful procedure and afterwards the video is analysed using the FLACC score. Each category is scored on a 0-2 scale (5 categories) which results in a total score of 0 (no pain) -10 (severe pain).

SECONDARY OUTCOMES:
adverse events of nitrous oxide 70% versus nitrous oxide 70% combined with fentanyl intranasal | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Seiler, Principal Investigator — University Children's Hospital of Zurich
Locations (1):
- Children's Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seiler M, Staubli G, Landolt MA. Combined nitrous oxide 70% with intranasal fentanyl for procedural analgosedation in children: a prospective, randomised, double-blind, placebo-controlled trial. Emerg Med J. 2019 Mar;36(3):142-147. doi: 10.1136/emermed-2018-207892. Epub 2019 Jan 10. PMID 30630844